CLINICAL TRIAL: NCT03790137
Title: An Open-Label Treatment of ZX008 (Fenfluramine Hydrochloride) in Pediatric and Adult Epilepsy Patients (Ages 4-25) With Sunflower Syndrome.
Brief Title: Treatment of Sunflower Syndrome With ZX008 (Fenfluramine Hydrochloride) in Children and Young Adults (Ages 4-25).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Elizabeth Anne Thiele (Other)
Collaborators: Zogenix International Limited, Inc., a subsidiary of Zogenix, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Elizabeth Anne Thiele, Director, Pediatric Epilepsy Program, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12112018
Record Dates: First submitted 2018-12-12; First posted 2018-12-31 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Photosensitive Epilepsy
Keywords: Sunflower Syndrome; Epilepsy
MeSH Terms: conditions — Epilepsy, Reflex; Epilepsy | interventions — Fenfluramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): The treatment group will include approximately 20 pediatric and young adult patients (ages 4-25 years) seen by Elizabeth A. Thiele, M.D., Ph.D. at MGH's Pediatric Epilepsy Clinic. Subjects will be treated on an outpatient basis and will not require hospital admission. The treatment group will receive the investigational new drug, Fenfluramine Hydrochloride for approximately 4 months. Patients that benefit from this treatment will remain on medication through an extension phase of the study.
  Interventions: Drug: Fenfluramine Hydrochloride

INTERVENTIONS:
Drug: Fenfluramine Hydrochloride — Fenfluramine Hydrochloride will be supplied to the treatment group as an oral solution in a concentration of 2.5 mg/mL. Subjects will receive their daily dose of Fenfluramine Hydrochloride in two doses (one in the morning and one in the evening). After a four week baseline, subjects that meet enrollment criteria will enter a titration period. The starting dose will be 0.2 mg/kg/day for the first 14 days. The dose will be increased every 2 weeks as tolerated by 0.2 mg/kg/day, to a maximum dose of 0.7 mg/kg/day, or a total maximum dose of 26 mg/day. The subject will remain on a dose of 0.7 mg/kg/day, 26 mg/day, or maximum tolerated daily dose through the end of the core study period.
  Other Names: ZX008

SUMMARY:
Sunflower Syndrome (also referred to as Self-induced Photosensitive Epilepsy) is a rare epileptic disorder characterized by a distinctive seizure that manifests itself in a highly stereotyped physical behavior. Seizure types associated with Sunflower Syndrome include absence seizures and generalized tonic-clonic seizures. Individuals with Sunflower Syndrome obsessively seek out a light source, stare at the light source, and wave one hand in front of their eye(s). Electroencephalogram (EEG) features include generalized spike and wave discharges interictally, and typically strong photoparoxysmal response during photic stimulation.

Currently, Sunflower syndrome is poorly characterized in medical literature and is often misunderstood at the clinical level. The name self-induced photosensitive epilepsy may be a misnomer as research concerning the neurochemical and neuropsychological pathways cannot conclusively determine that it is self-induced (conscious behavior) as the name implies. Although some reports have concluded that the hand waiving induces the seizure, these findings are not consistent throughout scientific literature. In fact, an EEG report found that the seizures can begin simultaneously with the hand waving. This suggests that the hand waving may in fact be part of the seizure, not the cause.

There are no treatments specifically approved for the treatment of Sunflower Syndrome in the United States. Broad spectrum anticonvulsant medications, including sodium valproate, lamotrigine, levetiracetam, and clobazam, have not shown full efficacy in seizure prevention in patients with Sunflower Syndrome. Accordingly, there remains a significant unmet need for an approved treatment for children and adults with Sunflower Syndrome.

Because this epilepsy typically does not respond to anticonvulsant medications, and because Aicardi described the successful treatment with fenfluramine of at least one child with this syndrome, the investigators of this study will investigate if fenfluramine is an effective, safe and well tolerated treatment for Sunflower Syndrome.

The primary objective of this study is to determine the efficacy of ZX008 on seizure frequency in children and young adults with Sunflower Syndrome. The goal of treatment is to provide a 30 percent or greater reduction of generalized tonic-clonic seizures and/or hand waving associated with absence seizures.

Secondary objectives of the study include evaluation of the effect of ZX008 (fenfluramine hydrochloride) on EEG patterns and quality of life. Patients with Sunflower Syndrome often experience low self-esteem, bullying due to the unusual motor movements associated with their seizures, school performance issues, anxiety, and depression.

The study population will include pediatric and young adult patients seen by Elizabeth A. Thiele, M.D., Ph.D. at MGH's Pediatric Epilepsy Clinic who were identified as candidates. The Principal Investigator (PI) will follow up to 20 patients with Sunflower Syndrome who will be taking ZX008.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or non-pregnant, non-lactating female, age 4 to 25 years, inclusive as of the day of the screening visit. Female subjects of childbearing potential must have a negative serum pregnancy test at screening. Subjects of childbearing or child-fathering potential must be willing to use medically acceptable forms of birth control, which includes abstinence, while in this study and for 90 days after the last dose of study drug.
* Subjects must have a diagnosis of Sunflower Syndrome, where seizures are not completely controlled by their current treatment plan.
* Subjects must experience seizures including absence seizures and/or generalized tonic-clonic seizures which involve seeking out a light source, staring at the light source, and waving one hand in front of their eye(s). Subject's must experience an average of 6 hand waving associated with absence seizures and/or generalized tonic-clonic seizures per week.
* Evidence of EEG in the medical history that shows generalized spike and wave discharges between seizures and a strong photoparoxysmal response during photic stimulation. Acceptable evidence includes a copy of the EEG trace, EEG report, or physician note that appropriately describes the EEG findings.
* All medications or interventions for epilepsy must be stable for at least 4 weeks prior to screening and are expected to remain stable until Month 3.
* Subject and/or parent/guardian has been informed of the nature of the study and informed consent has been obtained from the subject and/or legally responsible parent/guardian.
* Subject has provided assent in accordance with Institutional Review Board (IRB)/Ethics Committee requirements, if capable.
* Subjects parent/caregiver is willing and able to be compliant with diary completion, visit schedule, and study drug accountability.

Exclusion Criteria:

* Subject has a known hypersensitivity to fenfluramine hydrochloride or any other ingredients in the investigational drug,
* Subject's etiology of seizures is a degenerative neurological disease.
* Subject is pregnant.
* Subject is not willing to comply with a method of birth control acceptable to the PI during the study and for 90 days following completion of the study.
* Subject is breastfeeding.
* Subject has a history of drug or alcohol abuse.
* Subject has pulmonary arterial hypertension.
* Subject has current or past history of cardiovascular or cerebrovascular disease, such as cardiac valvulopathy, myocardial infarction or stroke, or clinically significant structural cardiac abnormality, including but not limited to mitral valve prolapse, atrial or ventricular septal defects, patent ductus arteriosis, and patent foramen ovale with reversal of shunt. (note: bicuspid valve is not considered exclusionary, but may be associated with the following diseases, which are exclusionary: coarctation of the aorta, Turner syndrome, supravalvular aortic stenosis, subvalvular aortic stenosis, patent ductus arteriosus, Sinus of Valsalva aneurysm, ventricular septal defect, Shone's complex, ascending aortic aneurysm, Loeys-Dietz syndrome, ACTA2 mutation familial thoracic aortic aneurysm syndrome, and MAT2A mutation familial thoracic aortic aneurysm syndrome).
* Subject has current or recent history of anorexia nervosa, bulimia, or depression within the prior year that required medical treatment or psychological treatment for a duration greater than 1 month.
* Subject has a current or past history of glaucoma.
* Subject has had an anoxic episode requiring resuscitation within 6 months of the screening visit.
* Subject has moderate or severe hepatic impairment. Asymptomatic subjects with mild hepatic impairment (elevated liver enzymes < 3x upper limit of normal (ULN) and/or elevated bilirubin <2x ULN) may be entered into the study after review and approval by the Medical Monitor in conjunction with the sponsor, in consideration of comorbidities and concomitant medications.
* Subject has severe renal impairment (estimated glomerular filtration rate <30mL/min/1.73m2)
* Subject is receiving concomitant therapy with: centrally-acting anorectic agents; monoamine-oxidase inhibitors; any centrally-acting compound with clinically appreciable amount of serotonin agonist or antagonist properties, including serotonin reuptake inhibition; other centrally-acting noradrenergic agonists, including atomoxetine; or cyproheptadine. (Note: Short-term medication requirements for prohibited medications will be handled on a per case basis by the medical monitor.)
* Subject has positive result (as defined in the laboratory manual) on urine tetrahydrocannabinol (THC) Panel or whole blood cannabidiol (CBD) at the screening visit.
* Subject has been taking felbamate for less than 1 year prior to screening and/or does not have stable liver function and hematology laboratory tests, and/or the dose has not been stable for at least 60 days prior to the screening visit.
* Subject is known to be human immunodeficiency virus (HIV) positive.
* Subject is known to have active viral hepatitis (B or C).
* Subject is currently receiving an investigational medicinal product.
* Subject has participated in another clinical trial within the past 30 days (calculated from that study's last scheduled visit). Participation in non-treatment trials will be reviewed by the medical monitor.
* Subject is at imminent risk of self-harm or harm to others, in the investigator's opinion.
* Subject is unwilling or unable to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions.
* Subject is institutionalized in a general nursing home (i.e., in a facility that does not provide skilled epilepsy care).-Subject does not have a reliable caregiver who can provide seizure diary information throughout the study.
* Subject has a clinically significant condition, or has had clinically relevant symptoms or a clinically significant illness in the 4 weeks prior to the Screening Visit, other than epilepsy, that would negatively impact study participation, collection of study data, or pose a risk to the subject.

Ages: 4 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2024-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Thiele, M.D., Ph.D., Principal Investigator — Director, Pediatric Epilepsy Program
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be made available to other researchers.

REFERENCES:
- [Background] Aicardi J, Gastaut H. Treatment of self-induced photosensitive epilepsy with fenfluramine. N Engl J Med. 1985 Nov 28;313(22):1419. doi: 10.1056/NEJM198511283132218. No abstract available. PMID 3932858
- [Background] Ames FR. "Self-induction" in photosensitive epilepsy. Brain. 1971;94(4):781-98. doi: 10.1093/brain/94.4.781. No abstract available. PMID 5132972
- [Background] Ames FR, Saffer D. The sunflower syndrome. A new look at "self-induced" photosensitive epilepsy. J Neurol Sci. 1983 Apr;59(1):1-11. doi: 10.1016/0022-510x(83)90076-x. PMID 6854340
- [Background] Belcastro V, Striano P. Self-induction seizures in sunflower epilepsy: a video-EEG report. Epileptic Disord. 2014 Mar;16(1):93-5. doi: 10.1684/epd.2014.0630. PMID 24556582
- [Background] Boel M, Casaer P. Add-on therapy of fenfluramine in intractable self-induced epilepsy. Neuropediatrics. 1996 Aug;27(4):171-3. doi: 10.1055/s-2007-973781. PMID 8892363
- [Background] Chieffo D, Battaglia D, Lettori D, Del Re M, Brogna C, Dravet C, Mercuri E, Guzzetta F. Neuropsychological development in children with Dravet syndrome. Epilepsy Res. 2011 Jun;95(1-2):86-93. doi: 10.1016/j.eplepsyres.2011.03.005. Epub 2011 Apr 6. PMID 21474289
- [Background] Fuller RW, Snoddy HD, Robertson DW. Mechanisms of effects of d-fenfluramine on brain serotonin metabolism in rats: uptake inhibition versus release. Pharmacol Biochem Behav. 1988 Jul;30(3):715-21. doi: 10.1016/0091-3057(88)90089-5. PMID 2463643
- [Background] LIVINGSTON S, TORRES IC. PHOTIC EPILEPSY: REPORT OF AN UNUSUAL CASE AND REVIEW OF THE LITERATURE. Clin Pediatr (Phila). 1964 May;3:304-7. doi: 10.1177/000992286400300511. No abstract available. PMID 14124883
- [Derived] Patel S, Geenen KR, Dowless D, Bruno PL, Thiele EA. Follow-up to low-dose fenfluramine for Sunflower syndrome: A non-randomized controlled trial. Dev Med Child Neurol. 2023 Jul;65(7):961-967. doi: 10.1111/dmcn.15492. Epub 2022 Dec 23. PMID 36562419
- See also: Zogenix Announces Positive Top-line Results from Pivotal Phase 3 — https://globenewswire.com/news-release/2017/09/29/1134829/0/en/Zogenix-Announces-Positive-Top-line-Results-from-Pivotal-Phase-3-Clinical-Trial-of-ZX008-in-Dravet-Syndrome.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After signing consent and enrolling in the study, all patients underwent a baseline echocardiogram, as well as baseline labs. If there were abnormal findings, patients were excluded from participation due to concerns of cardiac toxicity with fenfluramine.
Groups:
- Treatment Group: The treatment group will include approximately 20 pediatric and young adult patients (ages 4-25 years) seen by Elizabeth A. Thiele, M.D., Ph.D. at MGH's Pediatric Epilepsy Clinic. Subjects will be treated on an outpatient basis and will not require hospital admission. The treatment group will undergo a one month baseline, and then will take the investigational new drug, fenfluramine, for at least 84 days (~3 months). They will remain on treatment beyond the core study if fenfluramine is deemed effective and well-tolerated.
  Fenfluramine: Fenfluramine will be supplied to the treatment group as an oral solution. Subjects will receive their daily dose of Fenfluramine in two doses (one in the morning and one in the evening). After a four week baseline, all subjects that meet enrollment criteria will enter a titration period. The starting dose will be 0.2 mg/kg/day for the first 14 days. The dose will be increased every 2 weeks as tolerated by 0.2 mg/kg/day, to a maximum dose of 0.7 mg/kg/day (total maximum dose: 26 mg/day). The subjects will remain on a maximum dose for the duration of the core study.
Period: Overall Study
Arm/Group | Treatment Group
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: The treatment group will include approximately 20 pediatric and young adult patients (ages 4-25 years) with Sunflower syndrome seen by Elizabeth A. Thiele, M.D., Ph.D. at MGH's Pediatric Epilepsy Clinic. Subjects will be treated on an outpatient basis and will not require hospital admission. The treatment group will receive the investigational new drug, Fenfluramine Hydrochloride during the core study and may proceed to an extension phase of the study if there is perceived benefit.
  Fenfluramine Hydrochloride: Fenfluramine Hydrochloride will be supplied to the treatment group as an oral solution in a concentration of 2.5 mg/mL. Subjects will receive their daily dose of Fenfluramine Hydrochloride in two doses (one in the morning and one in the evening). After a four week baseline, subjects that meet enrollment criteria will enter a titration period. The starting dose will be 0.2 mg/kg/day for the first 14 days. The dose will be increased every 2 weeks as tolerated by 0.2 mg/kg/day, to a maximum dose of 0.7 mg/kg/day, or a total maximum dose of 26 mg/day. The subject will remain on a dose of 0.7 mg/kg/day, 26 mg/day, or maximum tolerated daily dose for the duration of the core study.
Arm/Group | Treatment Group
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 11.9 [7 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: % Change in Frequency of Handwaving Episodes
Description: The number of handwaving episodes (seizures) per day were recorded on a seizure diary by either the subject or the parent of the subject. One handwaving episode was defined as the period starting from when the hand first came up toward the face, until there was a brief pause in waving. Subjects and their caregivers were instructed to record the total number of handwaving episodes each day during a one month baseline, and during the 3 month treatment period.
  The baseline seizure frequency was calculated as an average of the reported handwaving episodes per day during the baseline period. This number was compared to the average episodes per day for the final month of the study (month 3 of treatment with fenfluramine) for each patient. The median percent change in frequency of handwaving episodes across all patients is reported below.
Time Frame: Month 3
Population: One patient withdrew from the study 3 days after starting study medication. This patient developed a rash, which was not thought to be related to study medication. The patient chose not to challenge the drug at an allergists office, and instead withdrew from the study. The other 19 patients completed the core study, but only 17 provided analyzable seizure data.
Measure: Median (95% Confidence Interval); unit: % change in hand waving episodes
Groups:
- Treatment Group: The treatment group will include approximately 20 pediatric and young adult patients (ages 4-25 years) with Sunflower syndrome.
Arm/Group | Treatment Group
Number analyzed (Participants) | 17
% change in hand waving episodes | -66.2 [-78.7 to -31.3]
Statistical Analysis 1: Comparison: Treatment Group; Test type: Other — The frequency of HWE for each patient was reported as episodes/day, as determined by dividing the total number of seizures experienced over a given time period by the number of days for which seizures were recorded. Paired t-tests were performed to compare each patient's baseline seizure frequency to their seizure frequency in the last month of treatment. Change in seizure frequency is reported as percent change from baseline. An alpha of 0.05 was used for statistical significance; p < 0.001, t-test, 1 sided

2. Primary Outcome: Change in Frequency of Generalized Tonic-clonic Seizures
Description: Daily seizure logs will be maintained by either the subject or the parent of the subject and used to calculate seizure frequency. Frequency of Generalized Tonic-clonic seizures was recorded as an average number of seizures/day. The average number of tonic-clonic seizures per day during the baseline period was compared to the average number of tonic-clonic seizures per day during the final month (month 3) for each patient that had experienced at least one tonic-clonic seizure in their lifetime.
Time Frame: Month 3
Population: 10 of the 20 patients reported having a generalized tonic-clonic seizure at some point in their lives.
Measure: Mean (Full Range); unit: tonic-clonic seizures/day
Arm/Group | Treatment Group
Number analyzed (Participants) | 10
tonic-clonic seizures/day | 0 [0 to 0]

3. Secondary Outcome: Change in Spike Frequency on EEG
Description: The investigators will read and interpret pre-drug (baseline) and post-drug EEGs (month 3 of core study) for the first 9 patients. The average number of spikes/hour across these patients will be reported for both pre- and post-treatment EEGs.
Time Frame: Month 3
Population: The investigators read and interpreted pre-drug and post-drug EEGs for the first 9 patients that completed the core study. The remaining 10 patients did not undergo EEGs as part of this study, due to safety concerns during the COVID-19 pandemic.
Measure: Mean (Full Range); unit: spikes/hour
Arm/Group | Treatment Group
Number analyzed (Participants) | 9
spikes/hour
  Pre-Treatment | 73.9 [0 to 277.2]
  Post-Treatment | 50.4 [0 to 187.2]

4. Secondary Outcome: Number of Patients That Experienced a Photoparoxysmal Response on EEG
Description: The investigators will read and interpret pre- (baseline) and post-treatment (month 3) EEGs. The number of patients that experienced a photoparoxysmal response during the EEGs will be reported.
Time Frame: Month 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 9
Participants
  Baseline EEG (pre-treatment) | 5
  Month 3 EEG (post-treatment) | 3

5. Secondary Outcome: Changes in Cognitive Functioning Determined by the Weschler Abbreviated Scale of Intelligence (WASI-II Subtests)
Description: The Weschler Abbreviated Scale of Intelligence (WASI-II subtests) will be administered to the first 10 patients at baseline and 84 days after the start of the first dose of study drug. Results of these cognitive tests will be compared between baseline and 84 days post initial dose.
  The WASI-II measures cognitive functioning through 2 subtests, vocabulary and matrix reasoning. The raw scores on these subtests are combined to give a composite full-scale IQ (FSIQ) that is scaled to an average of 100 and standard deviation of 15.
  Maximum raw scores for the subtests are as follows (higher values are considered better and minimum score on each is 0).
  Vocabulary:
  ages 7-11: 47 ages 12-14: 53 ages 15-25: 59
  Matrix Reasoning:
  ages 6-8: 24 ages 9-25: 30
Time Frame: Month 3 (~84 days after the first dose of fenfluramine.)
Population: 9 of the first 10 patients completed the core study. The second 10 patients did not undergo neuropsychological testing as part of this study due to safety concerns during the COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 9
score on a scale
  Baseline | 97.89 (13.53)
  Month 3 | 106.22 (11.64)

6. Secondary Outcome: Changes in Cognitive Functioning Determined by the Weschler Intelligence Scale for Children (WISC-V) -Processing Speed Subtests.
Description: The Weschler Intelligence Scale for Children (WISC-V) -Processing Speed subtests will be administered at baseline and 84 days after the start of the first dose of study drug (Month 3; visit 5). Results of these cognitive tests will be compared between baseline and 84 days post initial dose.
  Raw scores for the coding and symbol search subtests will be used to evaluate processing speed. The maximum raw scores are as follows (the minimum score is 0 and higher scores are considered better).
  Coding:
  ages 6-7: 65 ages 8-16: 119
  Symbol search:
  ages 6-7: 45 ages 8-16: 60
Time Frame: Month 3 (approximately 84 days after the first dose of fenfluramine)
Population: 9 of the first 10 patients underwent neuropsychological testing as part of the core study. The remaining patients did not undergo this testing due to safety concerns during the COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 9
score on a scale
  Baseline | 89.63 (9.12)
  Month 3 | 92.14 (10.48)

7. Secondary Outcome: Changes in Quality of Life Determined by the Quality of Life in Childhood Epilepsy Questionnaire(QOLCE-16)
Description: The Quality of Life in Childhood Epilepsy Questionnaire will be administered at baseline, and 84 days after the first dose (Month 3; visit 5). This questionnaire assesses mood, social relationships, and behaviors. Results will be compared.
  The QOLCE assesses quality of life across 4 domains of functioning: cognitive, emotional, social and physical. Scores range from 0-100. Composite scores are calculated as a mean across all measures.
Time Frame: Month 3 (approximately 84 days after first dose of fenfluramine)
Population: 8 of the first 9 patients completed this testing as part of the core study. The remaining patients did not undergo this testing due to safety concerns during the COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 8
score on a scale
  Baseline | 60.41 (18.88)
  Month 3 | 60.76 (17.48)

8. Secondary Outcome: Changes in Executive Functioning Determined by The Behavioral Rating Inventory of Executive Function (BRIEF) Questionnaire.
Description: The Behavioral Rating Inventory of Executive Function (BRIEF) questionnaire will be administered at baseline, and 84 days after the first dose of fenfluramine (Month 3; Visit 5). This questionnaire assesses executive function across 8 clinical scales:
  1. Inhibit
  2. Shift
  3. Emotional Control
  4. Initiate
  5. Working Memory
  6. Plan/Organize
  7. Organization of Materials
  8. Monitor
  Item level scores are rated on a 3 point Likert Scale from 1-3:
  1. Never
  2. Sometimes
  3. Often
  The Global Executive Composite (GEC) score is the total score of all 8 clinical subscales. The item scores are summed for each scale and raw scores are converted to Tscores. The mean of the GEC score will be reported.
  T scores from 60 to 64 are considered mildly elevated. T scores from 65 to 69 are considered potentially clinically elevated. T scores at or above 70 are considered clinically elevated.
Time Frame: Month 3 (approximately 84 days after the first dose of fenfluramine)
Population: 7 of the first 9 patients provided pre- and post-treatment responses to the BRIEF questionnaire. The remaining patients did not undergo this testing due to safety concerns during the COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Treatment Group
Number analyzed (Participants) | 7
T Score
  Baseline Score | 61.29 (13.62)
  Month 3 Score | 58.50 (15.84)

9. Secondary Outcome: Changes in Self-Concept Determined by The Beck Self Report Inventory.
Description: The Beck Self Report Inventory will be administered at baseline, and 84 days after the first dose (Month 3; Visit 5). This questionnaire assesses self-concept, depression, anxiety, anger and disruptive behavior through a 100-item self-report.
  The raw scores for subscales are calculated in the following manner:
  * Add scores from Items 1-20 for the total Beck Self Concept Inventory for Youth (BSCI-Y) score.
  * Add scores from Items 21-40 for the total Beck Anxiety Inventory for Youth (BAI-Y) score.
  * Add scores from Items 41-60 for the total Beck Depression Inventory for Youth (BDI-Y) score.
  * Add scores from Items 61-80 for the total Beck Anger Inventory for Youth (BANI-Y) score.
  * Add scores from Items 81-100 for the total Beck Disruptive Inventory for Youth (BDBI-Y) score.
  Raw scores will be translated into T-scores.
  T-scores for BYI are as follows:
  * 55 or less = average
  * 55-59 = mildly elevated
  * 60-69 = moderately elevated
  * 70+ = extremely elevated
Time Frame: Month 3 (approximately 84 days after first dose of fenfluramine)
Population: 7 of the first 9 patients provided pre- and post-treatment responses to the Beck Self Report Inventory. The remaining patients did not undergo this testing due to safety concerns during the COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Treatment Group
Number analyzed (Participants) | 7
T-Score
  Baseline Score | 44.43 (13.43)
  Month 3 Score | 52.88 (14.23)

10. Secondary Outcome: Changes in Anxiety Determined by the Beck Self Report Inventory
Description: as for outcome 9
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Treatment Group
Number analyzed (Participants) | 7
T score
  Baseline Score | 47.29 (8.20)
  Month 3 Score | 45.13 (5.91)

11. Secondary Outcome: Changes in Depression Determined by the Beck Self Report Inventory
Description: as for outcome 9
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Treatment Group
Number analyzed (Participants) | 7
T score
  Baseline Score | 49.29 (12.38)
  Month 3 Score | 47.13 (11.72)

12. Secondary Outcome: Changes in Anger Determined by the Beck Self Report Inventory
Description: as for outcome 9
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Treatment Group
Number analyzed (Participants) | 7
T score
  Baseline Score | 45.00 (7.87)
  Month 3 Score | 41.75 (5.52)

13. Secondary Outcome: Changes in Disruptive Behavior Determined by the Beck Self Report Inventory
Description: as for outcome 9
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Treatment Group
Number analyzed (Participants) | 7
T score
  Baseline Score | 44.14 (5.08)
  Month 3 Score | 43.50 (5.76)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between Baseline and Month 3 of the study (~84 days after the first dose of fenfluramine).
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 16/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=19)
Fatigue (General disorders) | 7
Reduced Appetite (General disorders) | 8
Nocturnal Enuresis (General disorders) | 2
Viral Illness (General disorders) | 4
Diarrhea (Gastrointestinal disorders) | 2
Shortness of Breath (General disorders) | 2
Chest Pain (General disorders) | 1
Seasonal Allergies (General disorders) | 2
Rhinorrhea (General disorders) | 1
irritability (General disorders) | 1
palilalia (General disorders) | 1
low serum calcium level (General disorders) | 1
acne exacerbation (Skin and subcutaneous tissue disorders) | 1
rash (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT03790137/Prot_001.pdf